CLINICAL TRIAL: NCT05078463
Title: Transdermal Microneedle Patch To Enhance Topical Anaesthesia Before Intravenous Line Insertion for Blood Transfusion In Paediatric Thalassemia Patients
Brief Title: Efficacy of Transdermal Microneedle Patch for Topical Anesthesia Enhancement in Paediatric Thalassemia Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Collaborators: Institue of Microengineering and Nanoelectronics (IMEN), Universiti Kebangsaan Malaysia (Unknown); Universiti Kebangsaan Malaysia Medical Molecular Biology Institute (UMBI) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UKM PPI/111/8/JEP-2021-578; PRGS/2/2020/TK05/UKM/01/1 (Other Grant/Funding Number: Ministry of Science Technology & Innovation, Malaysia)
Record Dates: First submitted 2021-09-20; First posted 2021-10-14 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Thalassemia in Children
Keywords: Microneedle; Maltose Microneedle; Thalassemia in Children; Paediatric Thalassemia; Transdermal microneedle patch; EMLA; Intravenous cannulation; Blood transfusion; Intravenous line insertion
MeSH Terms: interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: A Sham PVA-PET Patch that has the same size and structure as the maltose microneedle will be used. The participants, care providers and outcome assessors will not be able to distinguish between the maltose and sham patch due to their similar size and structure. One of the study investigators (Ooi Kai Shen) will not be masked since the person will be instituting the interventions. However, the study investigator (Ooi Kai Shen) is not one of the outcome assessors or care providers for the study participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention A: Microneedle with 1 Finger Tip Unit (FTU) EMLA for 30 minutes (Experimental): A Maltose Microneedle array patch (size: 1 cm x 1 cm) containing 36 microneedles (the height, base width and tip radius of each microneedle are 400 μm, 100 μm and 3 μm, respectively) with 1 mm needle gap in between will be firmly applied for 5 seconds against the pre-specified 1 cm x 1 cm grid (which will be the ideal site for intravenous cannulation for blood transfusion) on the dorsal surface of the hand. 1 Finger Tip Unit (FTU) of EMLA cream (containing an equal amount (25 mg) of lidocaine 2.5% and prilocaine 2.5%) (approximately 0.68g/cm2) will then be topically applied for 30 minutes on the same site of microneedle application. Intravenous cannulation will subsequently be carried out.
  Interventions: Device: Microneedle; Drug: 1 Finger Tip Unit (FTU) EMLA Cream (30-minute application time)
- Intervention B: Microneedle with 0.5 Finger Tip Unit (FTU) EMLA for 30 minutes (Experimental): A Maltose Microneedle array patch (size: 1 cm x 1 cm) containing 36 microneedles (the height, base width and tip radius of each microneedle are 400 μm, 100 μm and 3 μm, respectively) with 1 mm needle gap in between will be firmly applied for 5 seconds against the pre-specified 1 cm x 1 cm grid (which will be the ideal site for intravenous cannulation for blood transfusion) on the dorsal surface of the hand. 0.5 Finger Tip Unit (FTU) of EMLA cream containing an equal amount (25 mg) of lidocaine 2.5% and prilocaine 2.5% (dose: approximately 0.369 g/cm2) will then be topically applied for 30 minutes on the same site of microneedle application. Intravenous cannulation will subsequently be carried out.
  Interventions: Device: Microneedle; Drug: 0.5 Finger Tip Unit (FTU) EMLA (30-minute application time)
- Intervention C: Microneedle with 1 Finger Tip Units (FTUs) EMLA for 15 minutes (Experimental): A Maltose Microneedle array patch (size: 1 cm x 1 cm) containing 36 microneedles (the height, base width and tip radius of each microneedle are 400 μm, 100 μm and 3 μm, respectively) with1 mm needle gap in between will be firmly applied for 5 seconds against the pre-specified 1 cm x 1 cm grid (which will be the ideal site for intravenous cannulation for blood transfusion) on the dorsal surface of the hand. One (1) Finger Tip Unit (FTU) of EMLA cream (containing an equal amount (25 mg) of lidocaine 2.5% and prilocaine 2.5%) (approximately 0.68g/cm2) will then be topically applied for 15 minutes on the same site of microneedle application. Intravenous cannulation will subsequently be carried out.
  Interventions: Device: Microneedle; Drug: 1 Finger Tip Unit (FTU) EMLA (15-minute application time)
- Intervention D: 1 Finger Tip Unit (FTUs) EMLA only and PVA-containing PET Sham Patch (Sham Comparator): A Polyvinyl Alcohol (PVA)-containing Polyethylene Terephthalate (PET) Sham Patch of 1 cm x 1cm size will be applied for 5 seconds against the pre-specified 1 cm x 1 cm grid (which will be the ideal site for intravenous cannulation for blood transfusion) on the dorsal surface of the hand. One (1) Finger Tip Unit (FTU) of EMLA cream (containing an equal amount (25 mg) of lidocaine 2.5% and prilocaine 2.5%) (approximately 0.68g/cm2) will then be topically applied for 30 minutes on the same site of microneedle application. Intravenous cannulation will subsequently be carried out.
  Interventions: Drug: 1 Finger Tip Unit (FTU) EMLA Cream (30-minute application time); Device: Sham Patch

INTERVENTIONS:
Device: Microneedle — Maltose Microneedle Patch (Patch Size: 1 cm x 1 cm, 36 microneedles per patch, microneedle's height, base width and tip radius are 400 μm, 100 μm and 3 μm, respectively) will be firmly applied for 5 seconds on the 1 cm x 1 cm site for IV cannulation on the dorsal surface of the hand for blood transfusion, prior to EMLA cream application.
  Other Names: Maltose Microneedle Array Patch; Maltose Microneedle Patch
  Arms: Intervention A: Microneedle with 1 Finger Tip Unit (FTU) EMLA for 30 minutes; Intervention B: Microneedle with 0.5 Finger Tip Unit (FTU) EMLA for 30 minutes; Intervention C: Microneedle with 1 Finger Tip Units (FTUs) EMLA for 15 minutes
Drug: 1 Finger Tip Unit (FTU) EMLA Cream (30-minute application time) — 1 Finger Tip Units (FTU) EMLA applied for 30 minutes on the dorsal surface of the IV cannulated hand for blood transfusion
  Other Names: EMLA topical cream
  Arms: Intervention A: Microneedle with 1 Finger Tip Unit (FTU) EMLA for 30 minutes; Intervention D: 1 Finger Tip Unit (FTUs) EMLA only and PVA-containing PET Sham Patch
Drug: 1 Finger Tip Unit (FTU) EMLA (15-minute application time) — 1 Finger Tip Unit (FTU) EMLA applied for 15 minutes on the dorsal surface of the IV cannulated hand
  Other Names: EMLA topical cream
  Arms: Intervention C: Microneedle with 1 Finger Tip Units (FTUs) EMLA for 15 minutes
Drug: 0.5 Finger Tip Unit (FTU) EMLA (30-minute application time) — 0.5 Finger Tip Unit (FTU) EMLA applied for 30 minutes on the dorsal surface of the IV cannulated hand for blood transfusion
  Other Names: EMLA topical cream
  Arms: Intervention B: Microneedle with 0.5 Finger Tip Unit (FTU) EMLA for 30 minutes
Device: Sham Patch — A Polyvinyl Alcohol (PVA)-containing Polyethylene Terephthalate (PET) Sham Patch of a size of 1cm x 1cm will be applied for 5 seconds against the pre-specified 1 cm x 1 cm grid on the dorsal surface of the IV cannulated hand for blood transfusion.
  Other Names: Polyvinyl Alcohol (PVA)-containing Polyethylene Terephthalate (PET) Sham Patch
  Arms: Intervention D: 1 Finger Tip Unit (FTUs) EMLA only and PVA-containing PET Sham Patch

SUMMARY:
Microneedle (MN) is the mimic of a hypodermic needle, composed of hundreds of micron-sized, out-of-plane protrusions, typically arranged in arrays on a patch that can be applied onto the skin. MN can be fabricated from a variety of materials, preferably biocompatible polymers. Maltose, a natural carbohydrate, is a safe and biocompatible product that can be fabricated into MNs that are biodegradable and soluble within minutes. So far, maltose MN efficacy in enhancing the transdermal drug delivery (TDD) of topical anaesthetic agent such as Eutectic Mixture of Local Anesthetics (EMLA) and thus reducing the pain experienced by paediatric thalassemic patients requiring intravenous cannulation for regular blood transfusion has not been extensively studied. Therefore, the goals of this research are: 1) To compare the VAS score between thalassemic paediatric patients receiving EMLA before IV cannulation for blood transfusion and those receiving EMLA without microneedle application; 2) To compare the skin conductance algesimeter index between those receiving EMLA and microneedle and those receiving EMLA without microneedle application prior to intravenous (IV) cannulation for blood transfusion; 3) To evaluate the agreement between VAS score and the skin conductance algesimeter index obtained via PainMonitor™ machine.

DETAILED DESCRIPTION:
This is a prospective, phase II, randomized, double-blind (participants and care providers), cross-over, negative controlled trial.

Prior to the administration of intervention / control, relevant clinic-demographic profiles (age, gender, ethnicity, anthropometric measurements, presence of comorbidities, thalassemia types etc) will be recorded and entered in the case report forms (CRFs) that are specifically designed for this study.

This research study uses Eutectic Mixture of Local Anesthetics (EMLA) Cream (lidocaine 2.5% and prilocaine 2.5%) as the topical anaesthetic agent. EMLA Cream is a eutectic emulsion mixture of lidocaine and prilocaine at 1:1 ratio (i.e. each gram of EMLA cream contains lidocaine and prilocaine, 25 mg each). A eutectic mixture has a lower melting temperature than each constituent's melting temperature. The anaesthetic efficacy of EMLA cream will be assessed via pain induced by intravenous (IV) cannulation and the primary endpoint is the participant's VAS score measured after applying EMLA Cream (with and without MN application) for 15 and 30 minutes.

The window period given to EMLA Cream for its effect to work will be based on the usual clinical practice observation where it is usually applied for 30 minutes prior to IV catheterization. The rationale behind it is due to logistical issues and for the day care's operational convenience. Nevertheless, in a busy clinical setting, the application time is sometimes shortened to 15 minutes for slight anaesthetic effect. Thus, the study investigators postulate that, with the aid of microneedle, the time to onset of action for EMLA Cream could be greatly reduced, thus requiring less time for EMLA cream to achieve its maximal effects.

According to the routine hospital protocol, all study participants received their blood transfusion based on the Good Clinical Practice (GCP) guidelines. For each participant, the individual will be randomized to one of the 24 treatment sequences and there will be a minimum of 3-weeks washout period before administering the next intervention.

The investigator identified and drew a grid of 1cm × 1cm on the dorsum hand, which served as an ideal site for cannulation. The administrator of intervention (procedurist) will apply either 1 Finger Tip Units (FTUs) of EMLA Cream (approximately 0.68g/cm2) or 0.5 Finger Tip Unit (FTU) (approximately 0.369 g/cm2) over the preparation area. If the patient is subjected to MN patching at his/her visit, the MN patch will be applied by thumb force with the pillar handler pressed firmly against the dorsal hand surface for 5 seconds, mimicking a stamping action, to patch MN to the skin entirely before applying EMLA cream. Otherwise, an empty (i.e without MN) PVA-containing PET sham patch will be applied instead. Besides, the height-to-base ratio (4:1) used for MN will also optimally minimise its adverse effects (pain, redness), thus preserving the masking (blinding) of study participants from knowing the types of interventions received. The preparation area will be covered with an adhesive dressing ( 3M™Tegaderm™, Maplewood, Minnesota, USA) after EMLA cream application. After the allocated application time (15 or 30 minutes), the attending medical officer will set up the transfusion line with a 22-gauge hypodermic needle inserted into the dorsum hand. Throughout the process, the parents/guardians will be allowed to stay by the patient's side at all times.

After the intervention is given to the patients, the participants will be guided on the operating manual for a 10-points, 100mm VAS pain score. The participants will be presented with a ruler that contains 100-mm slots with "No Pain" written on the left side and "Worst Pain" on the opposite right side.

After each procedure, the children then will be asked to move and place the slider in the slot that accurately describes his/her pain at the following time points: 1) right after application of MN/ sham patch or before EMLA Cream application (baseline VAS score); 2) one minute after IV cannulation. The investigator will record the location of the slot where the slider is placed in (millimetres (mm), clearly printed on the ruler's backside) and this will be the participant's VAS score. Throughout the process, there will be a trained nurse standing by at the day-care to assist the verification of the pain scale and to aid the participants who require additional assistance.

Besides, before applying MN patch and EMLA Cream, the patients will be attached with the PainMonitor™ (Med-Storm Innovation AS, Oslo, Norway) device whereby the electrodes will be attached to the hypothenar eminence of the opposite hand not receiving the blood transfusion. The skin conductance peaks (in microSiemens (μS) and the average rise time (in microSiemens per second (μS/s)) will be recorded. Those parameters indicate the skin's sympathetic nerve block induced by the applied EMLA cream.

For skin conductance algesimeter index, the readings right after MN / sham patch application (baseline skin conductance algesimeter index score) and one minute IV cannulation will be obtained from the PainMonitor™ machine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged at least 6 to 17 years old
2. Patients requiring venous cannulation for blood transfusion

Exclusion Criteria:

1. Patients with a previous history of sensitization or allergy to EMLA cream
2. Patients with a previous history of allergy to materials used in the study (e.g. Polyvinyl Alcohol (PVA), Polyethylene Terephthalate (PET), Maltose, Electrodes and Plaster constituents)
3. Patients receiving other forms of analgesic agents within 24 hours prior to the cannulation procedures
4. Patients with generalized skin disorders / rash
5. Patients who are agitated or aggressive

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Score (VAS) | The measurements will be made at 1 minute after IV cannulation which will be inserted following EMLA (with or without microneedle) application
  VAS score is measured in a continuous scale (range 0-100). It is obtained using a Med-05-100 VAS Pain Scale ruler (Schlenker Enterprises Ltd, Lombard, USA) with 0-100 mm slider. It is measured based on the pain experienced on the IV cannulated hand for blood transfusion. Higher VAS score indicates greater intensity or degree of pain whilst lower VAS score indicates lesser pain intensity.
Skin Conductance Algesimeter Index | The measurements will be made at 1 minute after IV cannulation which will be inserted following EMLA (with our without microneedle) application
  The skin conductance peaks per second, measured in microSiemens per second (μS/s), is obtained using PainMonitor™ (Med-Storm Innovation AS, Oslo, Norway) device on the hypothenar eminence of the opposite hand not receiving blood transfusion. Higher skin conductance algesimeter index indicates greater pain intensity and lower values indicate lesser pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: FOOK-CHOE CHEAH, MD, MRCPCH, PhD, Principal Investigator — HOSPITAL CANSELOR TUANKU MUHRIZ, UNIVERSITI KEBANGSAAN MALAYSIA MEDICAL CENTER; AZRUL A HAMZAN, BSc, PhD, Principal Investigator — INSTITUTE OF MICROENGINEERING AND ELECTRONICS (IMEN), UKM; CHANG FU DEE, BSc, PhD, Principal Investigator — INSTITUTE OF MICROENGINEERING AND ELECTRONICS (IMEN), UKM; XIN YUN CHUA, BSc, Principal Investigator — HOSPITAL CANSELOR TUANKU MUHRIZ, UKM (UNIVERSITI KEBANGSAAN MALAYSIA MEDICAL CENTRE)
Locations (1):
- Hospital Canselor Tuanku Muhriz, Universiti Kebangsaan Malaysia (Ukm Medical Centre), Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual Participant Data (IPD) with information such as date of birth, hospital registration number and others that may lead to patient identification removed will be shared via Harvard Dataverse Repository after the end of trial and data collection.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The IPD will be made available to the public without any time frame limitation
Access Criteria: No access criteria are required. The data will be made available to the public, for all types of analyses for each study outcome measure, via the Harvard Dataverse repository, without requiring any access password or special access link.

REFERENCES:
- [Background] Waghule T, Singhvi G, Dubey SK, Pandey MM, Gupta G, Singh M, Dua K. Microneedles: A smart approach and increasing potential for transdermal drug delivery system. Biomed Pharmacother. 2019 Jan;109:1249-1258. doi: 10.1016/j.biopha.2018.10.078. Epub 2018 Nov 9. PMID 30551375
- [Background] Tucak A, Sirbubalo M, Hindija L, Rahic O, Hadziabdic J, Muhamedagic K, Cekic A, Vranic E. Microneedles: Characteristics, Materials, Production Methods and Commercial Development. Micromachines (Basel). 2020 Oct 27;11(11):961. doi: 10.3390/mi11110961. PMID 33121041
- [Background] Mooney K, McElnay JC, Donnelly RF. Children's views on microneedle use as an alternative to blood sampling for patient monitoring. Int J Pharm Pract. 2014 Oct;22(5):335-44. doi: 10.1111/ijpp.12081. Epub 2013 Dec 6. PMID 24308565
- [Background] Pires LR, Vinayakumar KB, Turos M, Miguel V, Gaspar J. A Perspective on Microneedle-Based Drug Delivery and Diagnostics in Paediatrics. J Pers Med. 2019 Nov 15;9(4):49. doi: 10.3390/jpm9040049. PMID 31731656
- [Background] Kim YC, Park JH, Prausnitz MR. Microneedles for drug and vaccine delivery. Adv Drug Deliv Rev. 2012 Nov;64(14):1547-68. doi: 10.1016/j.addr.2012.04.005. Epub 2012 May 1. PMID 22575858
- [Background] de Waard-van der Spek FB, van den Berg GM, Oranje AP. EMLA cream: an improved local anesthetic. Review of current literature. Pediatr Dermatol. 1992 Jun;9(2):126-31. doi: 10.1111/j.1525-1470.1992.tb01228.x. No abstract available. PMID 1603740
- [Background] Houck CS, Sethna NF. Transdermal analgesia with local anesthetics in children: review, update and future directions. Expert Rev Neurother. 2005 Sep;5(5):625-34. doi: 10.1586/14737175.5.5.625. PMID 16162086
- [Background] Duarah S, Sharma M, Wen J. Recent advances in microneedle-based drug delivery: Special emphasis on its use in paediatric population. Eur J Pharm Biopharm. 2019 Mar;136:48-69. doi: 10.1016/j.ejpb.2019.01.005. Epub 2019 Jan 8. PMID 30633972
- [Background] Ita K. Transdermal Delivery of Drugs with Microneedles-Potential and Challenges. Pharmaceutics. 2015 Jun 29;7(3):90-105. doi: 10.3390/pharmaceutics7030090. PMID 26131647
- [Background] Ali R, Mehta P, Arshad MS, Kucuk I, Chang MW, Ahmad Z. Transdermal Microneedles-A Materials Perspective. AAPS PharmSciTech. 2019 Dec 5;21(1):12. doi: 10.1208/s12249-019-1560-3. PMID 31807980
- [Background] Caffarel-Salvador E, Tuan-Mahmood TM, McElnay JC, McCarthy HO, Mooney K, Woolfson AD, Donnelly RF. Potential of hydrogel-forming and dissolving microneedles for use in paediatric populations. Int J Pharm. 2015 Jul 15;489(1-2):158-69. doi: 10.1016/j.ijpharm.2015.04.076. Epub 2015 May 1. PMID 25940042
- [Background] Kolli CS, Banga AK. Characterization of solid maltose microneedles and their use for transdermal delivery. Pharm Res. 2008 Jan;25(1):104-13. doi: 10.1007/s11095-007-9350-0. Epub 2007 Jun 28. PMID 17597381
- [Background] Taddio A, Ohlsson A, Einarson TR, Stevens B, Koren G. A systematic review of lidocaine-prilocaine cream (EMLA) in the treatment of acute pain in neonates. Pediatrics. 1998 Feb;101(2):E1. doi: 10.1542/peds.101.2.e1. PMID 9445511
- [Background] Beltramini A, Milojevic K, Pateron D. Pain Assessment in Newborns, Infants, and Children. Pediatr Ann. 2017 Oct 1;46(10):e387-e395. doi: 10.3928/19382359-20170921-03. PMID 29019634
- [Background] Storm H. Changes in skin conductance as a tool to monitor nociceptive stimulation and pain. Curr Opin Anaesthesiol. 2008 Dec;21(6):796-804. doi: 10.1097/ACO.0b013e3283183fe4. PMID 18997532
- [Background] Nayak A, Das DB, Vladisavljevic GT. Microneedle-assisted permeation of lidocaine carboxymethylcellulose with gelatine co-polymer hydrogel. Pharm Res. 2014 May;31(5):1170-84. doi: 10.1007/s11095-013-1240-z. Epub 2013 Nov 8. PMID 24203493
- [Background] Loizidou EZ, Inoue NT, Ashton-Barnett J, Barrow DA, Allender CJ. Evaluation of geometrical effects of microneedles on skin penetration by CT scan and finite element analysis. Eur J Pharm Biopharm. 2016 Oct;107:1-6. doi: 10.1016/j.ejpb.2016.06.023. Epub 2016 Jun 30. PMID 27373753
- [Background] Daly S, Claydon NCA, Newcombe RG, Seong J, Addy M, West NX. Randomised controlled trial of a microneedle patch with a topical anaesthetic for relieving the pain of dental injections. J Dent. 2021 Apr;107:103617. doi: 10.1016/j.jdent.2021.103617. Epub 2021 Feb 23. PMID 33636242

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/63/NCT05078463/Prot_SAP_ICF_001.pdf